CLINICAL TRIAL: NCT00511953
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo Controlled Study of the Pharmacokinetics (PK) and Pharmacodynamics (PD) of Gabapentin Extended Release (G-ER) Tablets in the Treatment of Vasomotor Symptoms in Postmenopausal Women
Brief Title: Study of Gabapentin Extended Release (G-ER) in the Treatment of Vasomotor (Hot Flashes/Hot Flushes) Symptoms in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Rekha Sathyanarayana, Depomed
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 81-0056
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Hot Flashes
Keywords: Hot flashes; Hot flushes; Postmenopausal symptoms
MeSH Terms: conditions — Hot Flashes | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin ER (Active Comparator): Active drug, Gabapentin extended release
  Interventions: Drug: Gabapentin Extended Release tablets; Drug: Gabapentin
- Sugar Pill (Placebo Comparator): Comparator arm is Placebo
  Interventions: Drug: Gabapentin Extended Release tablets; Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin Extended Release tablets — 1800mg
Drug: Gabapentin — 1800mg

SUMMARY:
Depomed's Gabapentin Extended Release is an investigational, extended release formulation of gabapentin that is being studied for the treatment of hot flashes in postmenopausal women.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to determine the optimal dose of Gabapentin ER in reducing the number and severity of hot flashes in postmenopausal women. Patients will be randomly assigned to Gabapentin ER or placebo, with a 1 in 4 chance of getting placebo. The total study investigational treatment duration after screening and baseline will be 13 weeks. The primary endpoint of the trial is to compare the number and severity of hot flashes during the investigational treatment compared to baseline. Sleep quality will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy, postmenopausal women who seek treatment for hot flashes.
2. Patients using hormone replacement therapy (HRT) must be willing to discontinue treatment.
3. Patients must be experiencing at least 7 moderate to severe hot flashes per day.
4. Patient must be willing to commit to 3 (optionally 4) overnight stays at the study site that will include frequent blood sampling.

Other inclusions apply.

Exclusion Criteria:

1. Patients with hypersensitivity to gabapentin.
2. Patients with severe chronic diarrhea, chronic constipation, uncontrolled irritable bowel syndrome (IBS) or unexplained weight loss.
3. Patients treated with estrogen pellets or injectable progestin drug therapy within 6 months.

Other exclusions apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Frequency of moderate to severe hot flashes reported during the corresponding 24- hour blood samples collection period | 24hrs
  PD end points are considered as primary outcomes of this study

SECONDARY OUTCOMES:
CGIC and PGIC evaluated prior to the start of 24- hour blood samples at week 6 and week 12 visits. | 12 wks
  Efficacy variables

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Burbank, California
  - DeLand, Florida
  - Port Orange, Florida
  - Shawnee, Kansas
  - Baltimore, Maryland
  - Hackensack, New Jersey
  - Greenville, South Carolina
  - San Antonio, Texas

REFERENCES:
- [Derived] Cowles VE, Gordi T, Hou SY. Steady-state pharmacokinetics of gabapentin after administration of a novel gastroretentive extended-release formulation in postmenopausal women with vasomotor symptoms. Clin Drug Investig. 2012 Sep 1;32(9):593-601. doi: 10.1007/BF03261914. PMID 22775354